CLINICAL TRIAL: NCT02672813
Title: Ultrasound Guided Pectoral Nerve I and II Blocks in Multimodal Analgesia for Breast Surgery: A Randomized Single Blinded Control Trial
Brief Title: Ultrasound Guided Pectoral Nerve I and II Blocks in Multimodal Analgesia for Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Anuranjan Ghimire, Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRC/521/015
Record Dates: First submitted 2016-01-28; First posted 2016-02-03 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Pain, Postoperative
Keywords: Pectoral nerve I and II blocks; Breast surgery; Ropivacaine; Postoperative opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pectoral Nerve I and II block (Experimental): Under Ultrasound guidance, Pectoral nerve I block is given for every breast surgery using 10ml of 0.25 % Ropivacaine ( without added preservatives). Similarly Pectoral nerve II block is also given using 20 ml of 0.25% Ropivacaine ( without added preservative) in same group of patient.
  Interventions: Procedure: Pectoral nerve I and II block
- No block (No Intervention): Pectoral nerve block is not given in this group of patients undergoing breast surgery

INTERVENTIONS:
Procedure: Pectoral nerve I and II block — Under Ultrasound guidance, Pectoral nerve I and II block is given for every breast surgery by using 10 and 20 ml of 0.25% Ropivacaine respectively
  Other Names: Pecs block
  Arms: Pectoral Nerve I and II block

SUMMARY:
The primary objective of this study is to access the effect of Pectoral nerve I and II blocks in breast surgery as measured by consumption of postoperative morphine or its equivalent.

DETAILED DESCRIPTION:
All patients in the study group and their relatives/attendants will be informed about the drugs, Pecs block and research methodology by the principal investigator during the pre-anaesthetic check up, in the evening before surgery. Informed and written consent will be obtained from the patient and/or his/her relatives. In order to assess pain, patient will be familiarized about the use of Numerical Rating Scale (NRS), in a language they can understand. (0 "as no pain at all" to 10 as "worst pain in life"). All of the patients will be premedicated with Tab diazepam 0.2mg/kg (not exceeding 10mg ) given orally night before surgery and in the morning of surgery.

On the day of surgery, after the patient arrives in the patient holding area in the operation theater, peripheral venous assess will be secured with 18G I.V cannula. In the operating room standard monitoring device will be attached to monitor Electrocardiograph ( ECG) , Pulse- oxymetry ( SpO2) , Non-invasive blood pressure ( NIBP), heart rate (HR) and End-tidal CO2 (Capnograph).

All patients will receive a standardized general anesthetic with multimodal analgesia. Preoxygenation will be done with 100% oxygen for three minutes. Induction will be done with loading dose of intravenous Fentanyl 1.5 mcg/kg and Propofol 1- 2 mg/kg and vecuronium 100mcg/kg. Airway will be secured by endotracheal intubation.

After induction of general anesthesia and before the start of surgery,ultrasound guided Pecs block will be performed by using 20-G Tuohy needle under all asceptic precautions. Images will be obtained using a Sonosite ultrasound machine. The probe will be placed at the mid clavicular level and angled inferolaterally,and then the axillary artery and vein will be located. The probe will then be moved laterally until pectoralis minor and serratus anterior are identified. The needle will be advanced in the tissue plane between Pectoralis major muscle (PMm) and Pectoralis minor muscle (Pmm) at the vicinity of pectoral branch of acromiothoracic artery and 10 ml of 0.25 % Ropivacine will be deposited. Similarly, 20ml of 0.25% Ropivacaine will be infiltrated in between Pmm and serratus anterior muscle at the level of third rib. (Blanco, R., Fajardo, M., Parras, M.T. 2006) Anesthesia will be maintained with isoflurane, oxygen, additional vecuronium and fentanyl. We will monitor Blood pressure, heart rate, SpO2, EtCO2, and ECG intraoperatively. During intraoperative period, 1gm of intravenous paracetomol will be given 15 minutes before the completion of surgery, over 15 minutes. Ondensatron (4mg IV) will be administered 15 minutes before the end of surgery as a prophylaxis for postoperative nausea and vomiting. Any episode of intraoperative hypotension (MAP lower than 65 mmHg) and bradycardia (heart rate < 50 bpm) will be treated with ephedrine 5 mg and atropine 0.4 mg IV respectively. On the completion of surgery,neuromuscular blockade will be reversed with 0.05 mg/kg of Neostigmine and 10mcg/kg of glycopyrrolate. The patient will then be extubated and transferred to postoperative recovery room.

In the postoperative recovery unit, blood pressure, pulse rate and oxygen saturation will be monitored for two hours. Assesment of pain scores at rest, coughing and on shoulder abuction along with postoperative nausea and vomiting (PONV) will be done in the postoperative recovery unit mmediately after patient will be transferred. If the patient has NRS of >3/10 at rest, intravenous morphine 2mg will be administered. If the pain is still not controlled, additional morphine of 2 mg can be given at 10 minute interval. PONV will be assessed by a categorical scale from 0 to 2. Intravenous ondensatron 4mg will be given if PONV scale is ≥1. If this proves to be ineffective, metoclopramide 10 mg will be administered. This rescue analgesia and antiemetic regimen will be followed for next 24 hours of surgery.

The patient will be transferred to ward on intravenous Ketorolac 30 mg every 8 hour and Ondensatron 4mg 8 hourly for 24 hours.

NRS for pain will be assessed immediately in postoperative recovery room and then at 2,4,8,12 and 24 hours of initial assessment.(on transfer to recovery). NRS will be calculated as 0 being "no pain" and 10 being "worst pain". NRS will also be assessed during coughing and abduction of ipsilateral shoulder in the at 0,2,8,12 and 24 hours of surgery. Similarly sedation score is also assessed at 0.2.4,8,12,and 24 hours after surgery ( 0 indicates the time of transfer to recovery and 2,4,8,12, and 24 meaning the time interval after 0 hour)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist ( ASA) Physical Status I, II
* Age between 16-65 Years
* Patients Undergoing breast surgery

Exclusion Criteria:

* Patient refusal
* Local infection
* Known hypersensitivity or any contraindications to study medication
* History of chronic pain
* Psychiatric illness
* Bilateral breast surgery
* Weight < 40 kg and > 100 kg

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Morphine consumption. | 24h
  Total amount of Morphine or its equivalent consumed by the patient in 24 hours following surgery is recorded

SECONDARY OUTCOMES:
Postoperative Numerical Rating scale (NRS) score for pain | 24 h
  NRS score for pain is used to assess the pain during rest , during coughing, and during abduction of ipsilateral shoulder within 24 hours following surgery at different time intervals
Satisfaction level | 24h
  Visual analog scale score for satisfaction level regarding the pain control after surgery is assessed at 24 hours of breast surgery
Nausea and Vomiting | 24h
  Number of patients who experience nausea and/or vomiting will be noted during the study
Local Anesthetic toxicity | 24h
  The occurrence of local anesthetic toxicity adverse reactions like pruritis, urticaria,headache, anxiety, confusion,tremors, tingling sensation, hypotension, cardiac arrhythmia, cardiac arrest, seizure will be noted and recorded during and after surgery.
sedation score | 24h
  5 point sedation scale is used to asses sedation within 24 hours at different time intervals ; where 0= alert, 1= arouses to voice, 2= arouses with gentle tactile stimulation, 3= arouses with vigorous tactile stimulation and 4= lack of responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Pokharel, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, Sunsari, Nepal